CLINICAL TRIAL: NCT04332692
Title: Acute Heart Failure - COngestion Discharge Evaluation. Évaluation de la Congestion à la Sortie d'Hospitalisation Pour Insuffisance Cardiaque aiguë.
Brief Title: Acute Heart Failure - COngestion Discharge Evaluation
Acronym: AHF-CODE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr. Nicolas GIRERD, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A03311-56
Record Dates: First submitted 2020-03-12; First posted 2020-04-03 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-03

CONDITIONS: Acute Heart Failure
Keywords: Acute Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients hospitalized for acute heart failure (Experimental): Patients hospitalized for acute heart failure will undergo the following evaluations:
  * Clinical examination focusing on congestion
  * Cardiac, pulmonary, peritoneal, jugular and renal venous Doppler ultrasounds
  * Blood sample retrieved for biological assessment and biobanking
  * Telephone follow-up
  Interventions: Procedure: Clinical examination centered on congestion; Procedure: Cardiac, pulmonary, peritoneal, jugular, renal Doppler ultrasounds and liver elastography; Procedure: Blood sample retrieved for biological assessment and biobanking; Procedure: Telephone follow-up; Behavioral: Kansas City Cardiomyopathy Questionnaire (KCCQ)

INTERVENTIONS:
Procedure: Clinical examination centered on congestion — Clinical examination centered on congestion (ASCEND, NYHA and Ambrosy Score) will be performed before discharge from hospital
Procedure: Cardiac, pulmonary, peritoneal, jugular, renal Doppler ultrasounds and liver elastography — Cardiac, pulmonary, peritoneal, jugular and renal Doppler ultrasounds and liver elastography will be performed before discharge from hospital
Procedure: Blood sample retrieved for biological assessment and biobanking — Blood sample retrieved for biological assessment and biobanking will be performed before discharge from hospital
Procedure: Telephone follow-up — Telephone follow-up will be performed 3, 12 and 24 months after discharge from hospital
Behavioral: Kansas City Cardiomyopathy Questionnaire (KCCQ) — Questionnaire centered on patient's quality of life at discharge and 3, 12 and 24 months after discharge

SUMMARY:
Acute heart failure (AHF) is a major public health problem, associated with a 40% risk of death or re-hospitalisation at 3 months. This risk is significantly increased by insufficient decongestion at the end of hospitalisation for AHF assessed by a standardised clinical score, a natriuretic peptide dosage or by cardiac and pulmonary ultrasound .

Adapting treatment according to lung congestion assessed by implantable devices (not reimbursed in France) improves the prognosis. However, due to the lack of a standardised congestion assessment, therapeutic adaptation in acute heart failure is currently empirical. The best multimodality approach to congestion evaluation is uncertain.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised for acute heart failure.
* Patients considered clinically discharging from hospitalisation for acute heart failure.
* Age ≥18 years
* Patients having received complete information regarding the study design and having signed their informed consent form.
* Patient affiliated to or beneficiary of a social security scheme.

Exclusion Criteria:

* Comorbidity for which the life expectancy is ≤ 3 months
* Dialysis patient (peritoneal dialysis or hemodialysis) or patients with glomerular filtration rate <15 ml/min/m2 at inclusion.
* History of lobectomy or pneumonectomy lung surgery
* Severe pulmonary or pleural pathology preventing reliable acquisition of lung ultrasound images: severe emphysema, chronic pleurisy, pulmonary fibrosis, etc.
* Pregnant woman, parturient or nursing mother
* Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* Adult person who is unable to give consent
* Person deprived of liberty by a judicial or administrative decision,
* Person subject to psychiatric care pursuant to Articles L. 3212-1 and L. 3213-1 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2028-05-20 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause death | 3 months after hospital discharge
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 2 and 3)
Rate of re-hospitalisation for acute heart failure | 3 months after hospital discharge
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 1 and 3)
Rate of day-hospital or in-home IV diuretics injection for acute HF | 3 months after hospital discharge
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 1 and 2)

SECONDARY OUTCOMES:
Rate of all-cause death | 3, 12 and 24 months after hospital discharge
Rate of re-hospitalisation for acute heart failure | 3,12 and 24 months after hospital discharge
Rate of day-hospital or in-home IV diuretics injection for acute HF | 3,12 and 24 months after hospital discharge
Rate of all-cause death | 12 and 24 months after hospital discharge
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF at 12 and 24 months following hospitalization (with outcome 8 and 9)
Rate of re-hospitalisation for acute heart failure | 12 and 24 months after hospital discharge
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF at 12 and 24 months following hospitalization (with outcome 7 and 9)
Rate of day-hospital or in-home IV diuretics injection for acute HF | 12 and 24 months after hospital discharge.
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF at 12 and 24 months following hospitalization (with outcome 7 and 8)
Rate of all-cause death | 3, 12 and 24 months after hospital discharge.
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 11 and 12)
Rate of hospitalization for acute heart failure | 3, 12 and 24 months after hospital discharge.
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 10 and 12)
Rate of day-hospital or in-home IV diuretics injection for acute HF | 3, 12 and 24 months after hospital discharge.
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 10 and 11)
NYHA (New York Heart Association) class measured | 3, 12 and 24 months after hospital discharge
Natriuretic peptides | within 24 months after hospital discharge.
  BNP or Nt-Pro BNP
Renal function assessed by glomerular filtration rate | within 24 months after hospital discharge.
Plasma volume | within 24 months after hospital discharge.
  calculated from haemoglobin and haematocrit value
Liver elastography value | At inclusion
  Measured with Fibroscan
Quality of life | At inclusion and 3, 6 and 24 months
  Assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, MD,PhD, Principal Investigator — CHRU of Nancy
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France